CLINICAL TRIAL: NCT00330226
Title: Naturalistic Prospective Follow-Up of Patients With Schizophrenia or Bipolar Disorders Receiving Atypical Antipsychotics and/or Mood Stabilizers
Brief Title: Efficacy and Safety of Psychopharmacotherapy in Patients With Schizophrenia or Bipolar Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Yong Min Ahn/Associate Professor, Seoul National University Hospital
Other Study IDs: KYS-2006-05318
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: schizophrenia; bipolar disorder; atypical antipsychotics; mood stabilizers; biological markers
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — regular lab tests for evaluating the changes in medical condition
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psychopharmacotherapy: patients under antipsychotic or mood stabilizer treatment

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of long-term psychopharmacotherapy in schizophrenia or bipolar disorder in terms of psychopathology and side effects.

DETAILED DESCRIPTION:
Schizophrenia and bipolar disorder are renowned for chronic and deteriorating course. Although atypical antipsychotics and mood stabilizers are widely used as treatment of choice for these illness based on acute efficacy and safety, long-term efficacy and safety of these agents are still open to debate. Prospective follow-up study in naturalistic condition may be a useful way of elucidating cons and pros of long-term psychopharmacotherapy.In this study, efficacy and various side effects of drugs will be measured, and the possibility of neurophysiological markers will be tested by serial measurements of electroencephalographic changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18-65 years of age.
* Patients must have a diagnosis of schizophrenia or bipolar disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
* Patients have not been received antipsychotics or mood stabilizers within the past 4 weeks prior to the study entry.
* Each patient must provide written informed consent after full explanation of study protocol, and authorized legal guardian must understand the nature of the study and must also give assent to study participation.

Exclusion Criteria:

* History of taking antipsychotics or mood stabilizers within past 4 weeks.
* History of DSM-IV substance dependence.
* Mental retardation (IQ < 70)or patients who are not able to understand the informed consent.
* Definite or suspected organic mental disorders.
* Female patients who are not able to maintain contraception during this study
* Laboratory abnormalities with clinical significance
* History of epilepsy or electroconvulsive therapy within the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with schizophrenia or bipolar disorder receiving pharmacotherapy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-01; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sik Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Angst F, Stassen HH, Clayton PJ, Angst J. Mortality of patients with mood disorders: follow-up over 34-38 years. J Affect Disord. 2002 Apr;68(2-3):167-81. doi: 10.1016/s0165-0327(01)00377-9. PMID 12063145
- [Background] Dunner DL. Safety and tolerability of emerging pharmacological treatments for bipolar disorder. Bipolar Disord. 2005 Aug;7(4):307-25. doi: 10.1111/j.1399-5618.2005.00235.x. PMID 16026484
- [Background] Kane JM. Treatment of schizophrenia. Schizophr Bull. 1987;13(1):133-56. doi: 10.1093/schbul/13.1.133. PMID 2885912
- [Background] Melkersson K, Dahl ML. Adverse metabolic effects associated with atypical antipsychotics: literature review and clinical implications. Drugs. 2004;64(7):701-23. doi: 10.2165/00003495-200464070-00003. PMID 15025545
- [Background] McGlashan TH. Early detection and intervention in schizophrenia: research. Schizophr Bull. 1996;22(2):327-45. doi: 10.1093/schbul/22.2.327. PMID 8782289
- [Background] Swann AC. Long-term treatment in bipolar disorder. J Clin Psychiatry. 2005;66 Suppl 1:7-12. PMID 15693746
- See also: Click here for the information about schizophrenia. — http://www.nlm.nih.gov/medlineplus/schizophrenia.html